CLINICAL TRIAL: NCT02034110
Title: A Phase II, Open-label, Study in Subjects With BRAF V600E-Mutated Rare Cancers With Several Histologies to Investigate the Clinical Efficacy and Safety of the Combination Therapy of Dabrafenib and Trametinib
Brief Title: Efficacy and Safety of the Combination Therapy of Dabrafenib and Trametinib in Subjects With BRAF V600E- Mutated Rare Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 117019; 2013-001705-87 (EudraCT Number); CDRB436X2201 (Other: Novartis); BRF117019 (Other: GlaxoSmithKline)
Record Dates: First submitted 2013-12-05; First posted 2014-01-13 (Estimated); Results first posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-07

CONDITIONS: Cancer
Keywords: solid tumors; anaplastic thyroid cancer (ATC); biliary tract cancer (BTC); gastrointestinal stromal tumor (GIST); low grade (WHO G1/G2) glioma (LGG); high grade (WHO G3/G4) glioma (HGG); non-seminomatous germ cell tumors (NSGCT)/non-germinomatous germ cell tumors (NGGCT); adenocarcinoma of the small intestine (ASI); hairy cell leukemia (HCL); multiple myeloma (MM); efficacy; safety; BRAF V600E mutation; Trametinib; Dabrafenib
MeSH Terms: conditions — Neoplasms; Thyroid Carcinoma, Anaplastic; Biliary Tract Neoplasms; Gastrointestinal Stromal Tumors; Glioma; Nonseminomatous germ cell tumor; Leukemia, Hairy Cell; Multiple Myeloma | interventions — dabrafenib; trametinib

STUDY DESIGN:
Intervention Model Description: 9 indications: anaplastic thyroid cancer (ATC), biliary tract cancer (BTC), gastrointestinal stromal tumor (GIST), low grade (WHO G1/G2) glioma (LGG), high grade (WHO G3/G4) glioma (HGG), non-seminomatous germ cell tumors (NSGCT)/non-germinomatous germ cell tumors (NGGCT), adenocarcinoma of the small intestine (ASI), hairy cell leukemia (HCL) and multiple myeloma (MM).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dabrafenib + Trametinib (Experimental): Subjects received Dabrafenib 150 mg twice daily orally plus Trametinib 2 mg once daily orally on a continuous basis. Dabrafenib was administered under fasted conditions, either 1 hour (hr) before or 2 hours (hrs) after a meal with approximately 200 mL of water with an interval of 12 hours. Trametinib was administered under fasted conditions, either 1 hr before or 2 hrs after a meal with approximately 200 mL of water. Subjects took their dose of Trametinib concurrently with the morning dose of Dabrafenib. A treatment cycle was 28 days in duration. Subjects continued treatment until an unacceptable toxicity, disease progression, or death occurs.
  Interventions: Drug: Dabrafenib; Drug: Trametinib

INTERVENTIONS:
Drug: Dabrafenib — A 150 mg twice daily capsule administered orally on a continuous basis.
  Other Names: DRB436; GSK2118436
Drug: Trametinib — A 2 mg once daily tablet administered orally on a continuous basis.
  Other Names: TMT212; GSK1120212

SUMMARY:
This was a Phase II, open-label, non-randomized, multi-center study of oral dabrafenib in combination with oral trametinib in subjects with rare cancers harboring the BRAF V600E mutation including anaplastic thyroid cancer (ATC), biliary tract cancer (BTC), gastrointestinal stromal tumor (GIST), low grade (WHO G1/G2) glioma (LGG), high grade (WHO G3/G4) glioma (HGG), non-seminomatous germ cell tumors (NSGCT) / non-germinomatous germ cell tumors (NGGCT), adenocarcinoma of the small intestine (ASI), hairy cell leukemia (HCL) and multiple myeloma (MM).

DETAILED DESCRIPTION:
This study was designed to determine the overall response rate (ORR) of oral Dabrafenib in combination with oral Trametinib in subjects with rare BRAF V600E mutated cancers. Subjects needed to have a fresh or frozen tumor tissue sample provided to confirm the BRAF V600E mutation status. Only subjects with histologically confirmed advanced disease and no available standard treatment options were eligible for enrollment. Subjects underwent screening assessments within 14 days (up to 35 days for ophthalmology exam, echocardiogram or disease assessments) prior to the start of treatment to determine their eligibility for enrollment in the study. All subjects enrolled received oral dabrafenib 150 mg bid in combination with oral trametinib 2 mg once daily. Subjects continued treatment until an unacceptable toxicity, disease progression, withdrawal of consent or death. Once a subject discontinued treatment, a post-treatment follow-up visit was conducted within 28 days (+ 7 days) after the last dose of study treatment(s). Extended follow-up visits were conducted every 4 weeks (+/- 7 days) for the first 6 months and then every 3 months (+/- 14 days) thereafter. A subject was considered to have discontinued the study if the subject was lost to follow-up or withdrew consent or another reason existed that prevented additional data from being collected on the subject. A subject was considered to have completed the study at the time of death.

For each histology, up to 25 patients were planned to be enrolled in each of the 9 primary analysis cohorts. A cohort could be closed or stopped early (prior to capping at 25 patients) for futility or efficacy. An uncapped expansion cohort was planned when a particular cohort was stopped early for efficacy. All planned histology cohorts enrolled at least one subject, with the exception of the germ cell tumor cohort. Enrolment in the study was closed in July 2018.

ELIGIBILITY:
Inclusion Criteria:

* Signed, written informed consent.
* Sex: male or female.
* Age: >=18 years of age at the time of providing informed consent.
* Eastern Cooperative Oncology Group (ECOG) performance status: 0, 1 or 2.
* Must have advanced disease and no standard treatment options as determined by locally/regionally available standards of care and treating physician's discretion
* Must have a a BRAF V600E mutation-positive tumor as confirmed by an approved local laboratory or a sponsor designated central reference laboratory. All subjects must provide an archived or fresh tumor sample (for solid tumors) or a fresh BM aspirate and peripheral blood sample (for HCL and MM) for confirmation testing of the BRAF V600E mutation by a sponsor designated central reference laboratory using a sponsor designated assay
* Able to swallow and retain orally administered medication. NOTE: Subject should not have any clinically significant gastrointestinal (GI) abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels. For example, subjects should have no more than 50% of the large intestine removed and no sign of malabsorption (i.e., diarrhea).NOTE: If clarification is needed as to whether a condition will significantly affect the absorption of study treatments, contact the GSK Medical Monitor.
* Female Subjects of Childbearing Potential: Subjects must have a negative serum pregnancy test within 7 days prior to the first dose of study treatment and agrees to use effective contraception, throughout the treatment period and for 4 months after the last dose of study treatment.
* French subjects: In France, a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category

Exclusion Criteria:

* Prior treatment with: BRAF and/or MEK inhibitor(s); anti-cancer therapy (e.g., chemotherapy with delayed toxicity, immunotherapy, biologic therapy or chemoradiation) within 21 days or prior nitrosourea or mitomycin C containing therapy within 42 days prior to enrollment and/or prior daily or weekly chemotherapy or biologic therapy without the potential for delayed toxicity within 14 days prior to enrolment or prior nvestigational drug(s) within 30 days or 5 half-lives, whichever is longer, prior to enrollment
* History of malignancy with confirmed activating RAS mutation at any time. Prospective RAS testing is not required. However, if the results of previous RAS testing are known, then those results must be used in assessing eligibility.
* Prior radiotherapy less than 14 days prior to enrollment, except for WHO Grade 1 4 glioma (radiotherapy is not permitted within 3 months prior to enrollment) and ATC (radiotherapy is not permitted within 7 days prior to enrollment). Treatment-related AEs must have resolved prior to enrollment.
* Prior major surgery less than 14 days prior to enrollment. Any surgery-related AE(s) must have resolved prior to enrollment
* Prior solid organ transplantation or allogenic stem cell transplantation (ASCT). However, previous autologous BM transplant (ABMT) or autologous peripheral blood stem cell transplant (PBSCT) is permitted.
* History of another malignancy. Subjects with another malignancy are eligible if: (a) disease-free for 3 years, or (b) have a history of completely resected non-melanoma skin cancer, and/or (c) have an indolent second malignancy(ies).
* Presence of brain metastases (except for subjects in the WHO Grade 1 or 2 or 3 or 4 glioma histology cohorts) that are symptomatic or untreated or not stable for >=3 months (must be documented by imaging) or requiring corticosteroids. Subjects on a stable dose of corticosteroids >14 days and have not required treatment with enzyme-inducing anticonvulsants for >30 days prior to enrollment can be enrolled with approval of the Medical Monitor
* Presence of symptomatic or untreated leptomeningeal or spinal cord compression. Subjects who have been previously treated for these conditions and have stable CNS disease (documented by consecutive imaging studies) for >60 days, are asymptomatic and currently not taking corticosteroids, or have been on a stable dose of corticosteroids for at least 30 days prior to enrollment, are permitted
* Presence of interstitial lung disease or pneumonitis
* Presence of any unresolved >=Grade 2 (per Common Terminology Criteria for Adverse Events [CTCAE] version 4.0) toxicity from previous anti-cancer therapy at the time of enrollment, except alopecia or Grade 2 anemia. Subjects with MM who have ≤Grade 2 peripheral neuropathy (per CTCAE v4.0) are permitted.
* Presence of any serious and/or unstable pre-existing medical disorder, psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures
* History of retinal vein occlusion
* Clinically significant GI abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels. For example, subjects should have no more than 50% of the large intestine removed and no sign of malabsorption (i.e., diarrhea)
* History or evidence of cardiovascular risk including any of the following: Acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within 6 months prior to enrolment; clinically significant uncontrolled arrhythmias; however, subjects with controlled atrial fibrillation for >30 days prior to enrollment are eligible; class II or higher congestive heart failure as defined by the New York Heart Association (NYHA) criteria; left ventricular ejection fraction (LVEF) below the institutional LLN. If a LLN does not exist at an institution, then use LVEF <50%; abnormal cardiac valve morphology (≥Grade 2) documented by ECHO; however, subjects with Grade 1 abnormalities (i.e., mild regurgitation/stenosis) may be entered on study but subjects with moderate valvular thickening should NOT be enrolled; corrected QT (QTc) interval for heart rate using Bazett-corrected QT interval (QTcB) >=480 msec; intracardiac defibrillator; treatment-refractory hypertension defined as a blood pressure (BP) >140/90 mmHg which may not be controlled by anti-hypertensive medication(s) and/or lifestyle modifications
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result within 3 months prior to first dose of study treatment. Subjects with positive Hepatitis C antibody due to prior exposure can be enrolled, only if a confirmatory negative Hepatitis C RNA polymerase chain reaction (PCR) test is obtained.
* Current use of prohibited medication(s) or requirement for prohibited medications during study as per the study protocol. Use of anticoagulants such as warfarin is permitted; however, international normalization ratio (INR) must be monitored according to local institutional practice.
* Clinically significant known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to study treatment, or excipients, or to dimethyl sulfoxide (structural component of dabrafenib).
* Pregnant, lactating or actively breastfeeding female subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2014-03-12 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (36):
- United States (7):
  - Novartis Investigative Site, Little Rock, Arkansas
  - Novartis Investigative Site, Santa Monica, California
  - Novartis Investigative Site, Bethesda, Maryland
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Houston, Texas
- Austria (4):
  - Novartis Investigative Site, Innsbruck
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
- Novartis Investigative Site, Jette, Belgium
- Novartis Investigative Site, Toronto, Ontario, Canada
- Novartis Investigative Site, Copenhagen, Denmark
- France (6):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Saint-Herblain
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Villejuif
- Germany (5):
  - Novartis Investigative Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Novartis Investigative Site, Heidelberg, Baden-Wurttemberg
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Hamburg
- Novartis Investigative Site, Milan, Lombardy, Italy
- Japan (2):
  - Novartis Investigative Site, Chiba
  - Novartis Investigative Site, Tokyo
- Netherlands (3):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Rotterdam
  - Novartis Investigative Site, Utrecht
- Novartis Investigative Site, Oslo, Norway
- Novartis Investigative Site, Seoul, South Korea
- Spain (2):
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Subbiah V, Burris HA 3rd, Kurzrock R. Revolutionizing cancer drug development: Harnessing the potential of basket trials. Cancer. 2024 Jan;130(2):186-200. doi: 10.1002/cncr.35085. Epub 2023 Nov 7. PMID 37934000
- [Derived] Hicks HM, Pozdeyev N, Sams SB, Pugazhenthi U, Bales ES, Hofmann MC, McKenna LR, Schweppe RE. Fibronectin Contributes to a BRAF Inhibitor-driven Invasive Phenotype in Thyroid Cancer through EGR1, Which Can Be Blocked by Inhibition of ERK1/2. Mol Cancer Res. 2023 Sep 1;21(9):867-880. doi: 10.1158/1541-7786.MCR-22-1031. PMID 37219859
- [Derived] Subbiah V, Kreitman RJ, Wainberg ZA, Gazzah A, Lassen U, Stein A, Wen PY, Dietrich S, de Jonge MJA, Blay JY, Italiano A, Yonemori K, Cho DC, de Vos FYFL, Moreau P, Fernandez EE, Schellens JHM, Zielinski CC, Redhu S, Boran A, Passos VQ, Ilankumaran P, Bang YJ. Dabrafenib plus trametinib in BRAFV600E-mutated rare cancers: the phase 2 ROAR trial. Nat Med. 2023 May;29(5):1103-1112. doi: 10.1038/s41591-023-02321-8. Epub 2023 Apr 14. PMID 37059834
- [Derived] Kreitman RJ, Moreau P, Ravandi F, Hutchings M, Gazzah A, Michallet AS, Wainberg ZA, Stein A, Dietrich S, de Jonge MJA, Willenbacher W, De Greve J, Arons E, Ilankumaran P, Burgess P, Gasal E, Subbiah V. Dabrafenib plus trametinib in patients with relapsed/refractory BRAF V600E mutation-positive hairy cell leukemia. Blood. 2023 Mar 2;141(9):996-1006. doi: 10.1182/blood.2021013658. PMID 36108341
- [Derived] Wen PY, Stein A, van den Bent M, De Greve J, Wick A, de Vos FYFL, von Bubnoff N, van Linde ME, Lai A, Prager GW, Campone M, Fasolo A, Lopez-Martin JA, Kim TM, Mason WP, Hofheinz RD, Blay JY, Cho DC, Gazzah A, Pouessel D, Yachnin J, Boran A, Burgess P, Ilankumaran P, Gasal E, Subbiah V. Dabrafenib plus trametinib in patients with BRAFV600E-mutant low-grade and high-grade glioma (ROAR): a multicentre, open-label, single-arm, phase 2, basket trial. Lancet Oncol. 2022 Jan;23(1):53-64. doi: 10.1016/S1470-2045(21)00578-7. Epub 2021 Nov 24. PMID 34838156
- [Derived] Subbiah V, Lassen U, Elez E, Italiano A, Curigliano G, Javle M, de Braud F, Prager GW, Greil R, Stein A, Fasolo A, Schellens JHM, Wen PY, Viele K, Boran AD, Gasal E, Burgess P, Ilankumaran P, Wainberg ZA. Dabrafenib plus trametinib in patients with BRAFV600E-mutated biliary tract cancer (ROAR): a phase 2, open-label, single-arm, multicentre basket trial. Lancet Oncol. 2020 Sep;21(9):1234-1243. doi: 10.1016/S1470-2045(20)30321-1. Epub 2020 Aug 17. PMID 32818466
- [Derived] Subbiah V, Kreitman RJ, Wainberg ZA, Cho JY, Schellens JHM, Soria JC, Wen PY, Zielinski C, Cabanillas ME, Urbanowitz G, Mookerjee B, Wang D, Rangwala F, Keam B. Dabrafenib and Trametinib Treatment in Patients With Locally Advanced or Metastatic BRAF V600-Mutant Anaplastic Thyroid Cancer. J Clin Oncol. 2018 Jan 1;36(1):7-13. doi: 10.1200/JCO.2017.73.6785. Epub 2017 Oct 26. PMID 29072975
- [Derived] Lee EQ, Ruland S, LeBoeuf NR, Wen PY, Santagata S. Successful Treatment of a Progressive BRAF V600E-Mutated Anaplastic Pleomorphic Xanthoastrocytoma With Vemurafenib Monotherapy. J Clin Oncol. 2016 Apr 1;34(10):e87-9. doi: 10.1200/JCO.2013.51.1766. Epub 2014 Aug 4. No abstract available. PMID 25092772

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 41 centers in 14 countries worldwide.
Pre-assignment Details: Subjects were enrolled into cohorts based on the type of histology. For each histology, up to 25 patients were planned to be enrolled. A cohort could be closed or stopped early (prior to capping at 25 patients) for futility or efficacy. An uncapped expansion cohort was planned when a particular cohort was stopped early for efficacy.
Groups:
- Anaplastic Thyroid Cancer (ATC); Biliary Tract Cancer (BTC); Gastrointestinal Stromal Tumor (GIST); Low Grade (WHO G1/G2) Glioma (LGG); High Grade (WHO G3/G4) Glioma (HGG); Adenocarcinoma of the Small Intestine (ASI); Hairy Cell Leukemia (HCL); Multiple Myeloma (MM): All subjects enrolled received oral dabrafenib 150 mg bid in combination with oral trametinib 2 mg once daily. Subjects continued treatment until an unacceptable toxicity, disease progression, or death.
Period: Overall Study
Arm/Group | Anaplastic Thyroid Cancer (ATC) | Biliary Tract Cancer (BTC) | Gastrointestinal Stromal Tumor (GIST) | Low Grade (WHO G1/G2) Glioma (LGG) | High Grade (WHO G3/G4) Glioma (HGG) | Adenocarcinoma of the Small Intestine (ASI) | Hairy Cell Leukemia (HCL) | Multiple Myeloma (MM)
Started (All enrolled participants were included in the Intent-to-treat (ITT), All-treated subjects (ATS) and ITT/Evaluable populations) | 36 | 43 | 1 | 13 | 45 | 3 | 55 | 10
Primary Analysis Cohort | 15 | 18 | 1 | 13 | 24 | 3 | 24 | 10
Expansion Cohort | 21 | 25 | 0 | 0 | 21 | 0 | 31 | 0
Completed | 24 | 34 | 1 | 4 | 28 | 3 | 8 | 9
Not Completed | 12 | 9 | 0 | 9 | 17 | 0 | 47 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 5 | 7 | 0 | 3 | 7 | 0 | 3 | 1
Not completed — Study closed by sponsor | 6 | 2 | 0 | 6 | 7 | 0 | 42 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anaplastic Thyroid Cancer (ATC) | Biliary Tract Cancer (BTC) | Gastrointestinal Stromal Tumor (GIST) | Low Grade (WHO G1/G2) Glioma (LGG) | High Grade (WHO G3/G4) Glioma (HGG) | Adenocarcinoma of the Small Intestine (ASI) | Hairy Cell Leukemia (HCL) | Multiple Myeloma (MM) | Total
Number analyzed (Participants) | 36 | 43 | 1 | 13 | 45 | 3 | 55 | 10 | 206
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.6 (9.53) | 57.0 (11.88) | 77.0 (NA) — Only one participant analyzed | 33.1 (11.51) | 41.9 (14.70) | 58.3 (3.21) | 64.8 (10.77) | 66.9 (6.89) | 57.1 (16.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 24 | 1 | 9 | 22 | 1 | 8 | 5 | 90
  Male | 16 | 19 | 0 | 4 | 23 | 2 | 47 | 5 | 116
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 4
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Asian - Central/South Asian Heritage | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian - East Asian Heritage | 11 | 1 | 0 | 0 | 4 | 0 | 0 | 1 | 17
  Asian - Japanese Heritage | 2 | 2 | 0 | 2 | 1 | 0 | 0 | 0 | 7
  Asian - South East Asian Heritage | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 4
  White - Arabic/North African Heritage | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 5
  White - White/Caucasian/European heritage | 17 | 39 | 1 | 10 | 32 | 2 | 48 | 8 | 157
  Missing | 2 | 0 | 0 | 0 | 2 | 0 | 6 | 0 | 10
ECOG Performance Status [Count of Participants; unit: Participants] — The Eastern Cooperative Oncology Group Performance Status (ECOG PS) score classifies participants according to their functional impairment, with scores ranging from 0 (fully active) to 5 (dead). ECOG PS: 0 = Fully active, able to carry on all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2 = ambulatory and capable of all self-care but unable to carry out any work activities, up and about more than 50% of waking hours
  Participants
    Grade 0 | 4 | 17 | 1 | 5 | 14 | 3 | 25 | 3 | 72
    Grade 1 | 30 | 24 | 0 | 7 | 24 | 0 | 27 | 6 | 118
    Grade 2 | 2 | 2 | 0 | 1 | 7 | 0 | 3 | 1 | 16

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) in the Anaplastic Thyroid Cancer (ATC) Cohort
Description: Overall Response Rate (ORR) was defined as the percentage of participants with a tumor response (complete response [CR], partial response [PR]) by investigator assessment as defined by RECIST v1.1. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: From study treatment start date until first documented complete response or partial response, assessed up to 78 months (cut-off date for FDA Submission = 14-Sep-20) and up to 92 months (cut-off date for end of study = 10-Dec-21)
Population: ITT/Evaluable population - Primary and expansion cohort combined
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Anaplastic Thyroid Cancer (ATC)
Number analyzed (Participants) | 36
Percentage of Participants
  Investigator assessment @ up to 78 months | 56 [38.1 to 72.1]
  Investigator assessment @ up to 92 months | 56 [38.1 to 72.1]
  Independent radiology review @ up to 78 months | 53 [35.5 to 69.6]
  Independent radiology review @ up to 92 months | 53 [35.5 to 69.6]

2. Primary Outcome: Overall Response Rate (ORR) in the Biliary Tract Cancer (BTC) Cohort
Description: as for outcome 1
Time Frame: as for outcome 1
Population: ITT/Evaluable population - Primary and expansion cohort combined
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Biliary Tract Cancer (BTC)
Number analyzed (Participants) | 43
Percentage of Participants
  Investigator assessment @ up to 78 months | 53 [37.7 to 68.8]
  Investigator assessment @ up to 92 months | 53 [37.7 to 68.8]
  Independent radiology review @ up to 78 months | 47 [31.2 to 62.3]
  Independent radiology review @ up to 92 months | 47 [31.2 to 62.3]

3. Primary Outcome: Overall Response Rate (ORR) in the Gastrointestinal Stromal Tumor (GIST) Cohort
Description: as for outcome 1
Time Frame: as for outcome 1
Population: ITT/Evaluable population - Primary and expansion cohort combined
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Gastrointestinal Stromal Tumor (GIST)
Number analyzed (Participants) | 1
Percentage of Participants
  Investigator assessment @ 78 months | 0 [NA to NA] — 95% Confidence Interval not determined as there are an insufficient number of participants with events.
  Investigator assessment @ 92 months | 0 [NA to NA] — 95% Confidence Interval not determined as there are an insufficient number of participants with events.

4. Primary Outcome: Overall Response Rate (ORR) in the Adenocarcinoma of the Small Intestine (ASI) Cohort
Description: as for outcome 1
Time Frame: as for outcome 1
Population: ITT/Evaluable population - Primary and expansion cohort combined
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Adenocarcinoma of the Small Intestine (ASI)
Number analyzed (Participants) | 3
Percentage of Participants
  Investigator assessment @ up to 78 months | 67 [9.4 to 99.2]
  Investigator assessment @ up to 92 months | 67 [9.4 to 99.2]

5. Primary Outcome: Overall Response Rate (ORR) in the Low Grade (WHO G1/G2) Glioma (LGG) Cohort
Description: Overall Response Rate (ORR) was defined as the percentage of participants with a tumor response (response assessment criteria (CR, PR, and minor response [MR]) WHO Grade 1 and 2 Glioma) by investigator assessment as defined by response assessment for neuro-oncology (RANO). Specifically, ORR = number of subjects with a confirmed overall response divided by the total number of subjects in the corresponding analysis population.
Time Frame: as for outcome 1
Population: ITT/Evaluable population - Primary analysis cohort
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Low Grade (WHO G1/G2) Glioma (LGG)
Number analyzed (Participants) | 13
Percentage of Participants
  Investigator assessment/Response rate @ up to 78 months | 69 [38.6 to 90.9]
  Investigator assessment/Response rate @ up to 92 months | 69 [38.6 to 90.9]
  Independent radiology review/Response rate @ up to 78 months | 69 [38.6 to 90.9]
  Independent radiology review/Response rate @ up to 92 months | 62 [31.6 to 86.1]

6. Primary Outcome: Overall Response Rate (ORR) in the High Grade (WHO G3/G4) Glioma (HGG) Cohort
Description: Overall Response Rate (ORR) was defined as the percentage of participants with a tumor response (updated response assessment criteria (CR, PR) WHO Grade 3 and 4 Glioma) by investigator assessment as defined by modified response assessment for neuro-oncology (RANO). Specifically, ORR = number of subjects with a confirmed overall response divided by the total number of subjects in the corresponding analysis population.
Time Frame: as for outcome 1
Population: ITT/Evaluable population - Primary and expansion cohort combined
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | High Grade (WHO G3/G4) Glioma (HGG)
Number analyzed (Participants) | 45
Percentage of Participants
  Investigator assessment @ up to 78 months | 33 [20.0 to 49.0]
  Investigator assessment @ up to 92 months | 33 [20.0 to 49.0]
  Independent radiology review @ up to 78 months | 31 [18.2 to 46.6]
  Independent radiology review @ up to 92 months | 31 [18.2 to 46.6]

7. Primary Outcome: Overall Response Rate (ORR) in the Hairy Cell Leukemia (HCL) Cohort
Description: Overall Response Rate (ORR) was defined as the percentage of participants with CR +/- minimal residual disease [MRD], PR by investigator assessment as defined by the Consensus Resolution Criteria adapted from the National Comprehensive Cancer Network (NCCN) guidelines. Specifically, ORR = number of subjects with a confirmed overall response divided by the total number of subjects in the corresponding analysis population.
Time Frame: as for outcome 1
Population: ITT/Evaluable population - Primary and expansion cohort combined
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Hairy Cell Leukemia (HCL)
Number analyzed (Participants) | 55
Percentage of Participants
  Investigator assessment @ up to 78 months | 89 [77.8 to 95.9]
  Investigator assessment @ up to 92 months | 89 [77.8 to 95.9]

8. Primary Outcome: Overall Response Rate (ORR) in the Multiple Myeloma (MM) Cohort
Description: Overall Response Rate (ORR) was defined as the percentage of participants with stringent complete response (sCR), CR, PR, very good partial response (VGPR) by investigator assessment as defined by the International Myeloma Working Group (IMWG) Uniform Response Criteria for Multiple Myeloma. Specifically, ORR = number of subjects with a confirmed overall response divided by the total number of subjects in the corresponding analysis population.
Time Frame: as for outcome 1
Population: ITT/Evaluable population - Primary analysis cohort
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Multiple Myeloma (MM)
Number analyzed (Participants) | 10
Percentage of Participants
  Investigator assessment @ up to 78 months | 50 [18.7 to 81.3]
  Investigator assessment @ up to 92 months | 50 [18.7 to 81.3]

9. Secondary Outcome: Duration of Response (DoR) in the Anaplastic Thyroid Cancer (ATC) Cohort
Description: For the subset of subjects who showed a confirmed response as defined for each cohort, Duration of Response (DoR) was defined as the time (in weeks) from first documented evidence of response (the first response prior to confirmation) until time of documented disease progression or death due to any cause, whichever was first. If the subject did not have a documented date of progression or death, DoR was censored at the date of the last adequate assessment.
Time Frame: From first documented evidence of response (the first response prior to confirmation) until time of documented disease progression or death due to any cause, whichever comes first, assessed up to 92 months (cut-off date for end of study = 10-Dec-21)
Population: ITT/Evaluable population - Primary and expansion cohorts combined. Only responders were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Anaplastic Thyroid Cancer (ATC)
Number analyzed (Participants) | 20
Weeks
  Investigator assessment | 62.4 [32.1 to NA] — Not estimable due to insufficient events observed.
  Independent radiology review | 59.1 [16.6 to 171.4]

10. Secondary Outcome: Duration of Response (DoR) in the Biliary Tract Cancer (BTC) Cohort
Description: as for outcome 9
Time Frame: as for outcome 9
Population: ITT/Evaluable population - Primary and expansion cohorts combined. Only responders were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Biliary Tract Cancer (BTC)
Number analyzed (Participants) | 23
Weeks
  Investigator assessment | 38.9 [24.3 to 59.4]
  Independent radiology review | 45.4 [20.1 to 64.9]

11. Secondary Outcome: Duration of Response (DoR) in the Adenocarcinoma of the Small Intestine (ASI) Cohort
Description: as for outcome 9
Time Frame: as for outcome 9
Population: ITT/Evaluable population - Primary analysis cohort. Only responders were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Adenocarcinoma of the Small Intestine (ASI)
Number analyzed (Participants) | 2
Weeks
  Investigator assessment | 33.4 [NA to NA] — Not estimable due to insufficient events observed.
  Independent radiology review | 32.8 [32.1 to NA] — Not estimable due to insufficient events observed.

12. Secondary Outcome: Duration of Response (DoR) in the Low Grade (WHO G1/G2) Glioma (LGG) Cohort
Description: as for outcome 9
Time Frame: as for outcome 9
Population: ITT/Evaluable population - Primary analysis cohort. Only responders were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Low Grade (WHO G1/G2) Glioma (LGG)
Number analyzed (Participants) | 9
Weeks
  Investigator assessment | NA [24.1 to NA] — Not estimable due to insufficient events observed
  Independent radiology review | 84.3 [16.4 to NA] — Not estimable due to insufficient events observed

13. Secondary Outcome: Duration of Response (DoR) in the High Grade (WHO G3/G4) Glioma (HGG) Cohort
Description: as for outcome 9
Time Frame: as for outcome 9
Population: ITT/Evaluable population - Primary and expansion cohorts combined. Only responders were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | High Grade (WHO G3/G4) Glioma (HGG)
Number analyzed (Participants) | 15
Weeks
  Investigator assessment | 135.7 [32.0 to 192.0]
  Independent radiology review | 59.3 [20.1 to 116.0]

14. Secondary Outcome: Duration of Response (DoR) in the Hairy Cell Leukemia (HCL) Cohort
Description: as for outcome 9
Time Frame: as for outcome 9
Population: ITT/Evaluable population - Primary and expansion cohorts combined. Only responders were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Hairy Cell Leukemia (HCL)
Number analyzed (Participants) | 49
Weeks | NA [NA to NA] — Not estimable due to insufficient events observed

15. Secondary Outcome: Duration of Response (DoR) in the Multiple Myeloma (MM) Cohort
Description: as for outcome 9
Time Frame: as for outcome 9
Population: ITT/Evaluable population - Primary analysis cohort. Only responders were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Multiple Myeloma (MM)
Number analyzed (Participants) | 5
Weeks | 48.1 [24.3 to NA] — Not estimable due to insufficient events observed

16. Secondary Outcome: Progression Free Survival (PFS) in the Anaplastic Thyroid Cancer (ATC) Cohort
Description: Progression Free Survival (PFS) was defined as the interval between the first dose of study treatment and earlier date of first radiologically documented progression or death due to any cause. If the subject did not have a documented date of progression or death, PFS was censored at the date of the last adequate assessment. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started.
Time Frame: From study treatment start date until date of radiographic progression or date of death from any cause, whichever comes first, assessed up to 92 months (cut-off date for end of study = 10-Dec-21)
Population: ITT/Evaluable population - Primary and expansion cohort combined
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Anaplastic Thyroid Cancer (ATC)
Number analyzed (Participants) | 36
Weeks
  Investigator assessment | 29.1 [20.3 to 59.9]
  Independent radiology review | 24.1 [16.1 to 56.0]

17. Secondary Outcome: Progression Free Survival (PFS) in the Biliary Tract Cancer (BTC) Cohort
Description: as for outcome 16
Time Frame: as for outcome 16
Population: ITT/Evaluable population - Primary and expansion cohort combined
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Biliary Tract Cancer (BTC)
Number analyzed (Participants) | 43
Weeks
  Investigator assessment | 39.0 [24.1 to 41.0]
  Independent radiology review | 32.6 [23.6 to 56.0]

18. Secondary Outcome: Progression Free Survival (PFS) in the Adenocarcinoma of the Small Intestine (ASI) Cohort
Description: as for outcome 16
Time Frame: as for outcome 16
Population: ITT/Evaluable population - Primary analysis cohort.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Adenocarcinoma of the Small Intestine (ASI)
Number analyzed (Participants) | 3
Weeks
  Investigator assessment | 41.3 [NA to NA] — Not estimable due to insufficient events observed
  Independent radiology review | 40.1 [4.1 to NA] — Not estimable due to insufficient events observed

19. Secondary Outcome: Progression Free Survival (PFS) in the Low Grade (WHO G1/G2) Glioma (LGG) Cohort
Description: Progression Free Survival (PFS) was defined as the interval between the first dose of study treatment and earlier date of first radiologically documented progression or death due to any cause. If the subject did not have a documented date of progression or death, PFS was censored at the date of the last adequate assessment.
Time Frame: as for outcome 16
Population: ITT/Evaluable population - Primary analysis cohort.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Low Grade (WHO G1/G2) Glioma (LGG)
Number analyzed (Participants) | 13
Weeks
  Investigator assessment | NA [32.1 to NA] — Not estimable due to insufficient events observed
  Independent radiology review | 40.1 [20.3 to 143.7]

20. Secondary Outcome: Progression Free Survival (PFS) in the High Grade (WHO G3/G4) Glioma (HGG) Cohort
Description: as for outcome 19
Time Frame: as for outcome 16
Population: ITT/Evaluable population - Primary and expansion cohort combined
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | High Grade (WHO G3/G4) Glioma (HGG)
Number analyzed (Participants) | 45
Weeks
  Investigator assessment | 24.0 [8.0 to 59.4]
  Independent radiology review | 19.7 [8.0 to 32.1]

21. Secondary Outcome: Progression Free Survival (PFS) in the Hairy Cell Leukemia (HCL) Cohort
Description: as for outcome 19
Time Frame: as for outcome 16
Population: ITT/Evaluable population - Primary and expansion cohort combined
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Hairy Cell Leukemia (HCL)
Number analyzed (Participants) | 55
Weeks | NA [NA to NA] — Not estimable due to insufficient events observed

22. Secondary Outcome: Progression Free Survival (PFS) in the Multiple Myeloma (MM) Cohort
Description: as for outcome 19
Time Frame: as for outcome 16
Population: ITT/Evaluable population - primary analysis cohort
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Multiple Myeloma (MM)
Number analyzed (Participants) | 10
Weeks | 27.5 [10.0 to 55.9]

23. Secondary Outcome: Overall Survival (OS) in the Anaplastic Thyroid Cancer (ATC) Cohort
Description: Overall Survival (OS) was defined as the time from first dose until death due to any cause. Censoring was performed using the date of last known contact for those who were alive at the time of analysis.
Time Frame: From study treatment start date until date of death from any cause, assessed up to 92 months (cut-off date for end of study = 10-Dec-21)
Population: ITT/Evaluable population - Primary and expansion cohort combined
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Anaplastic Thyroid Cancer (ATC)
Number analyzed (Participants) | 36
Weeks | 62.9 [29.6 to 100.9]

24. Secondary Outcome: Overall Survival (OS) in the Biliary Tract Cancer (BTC) Cohort
Description: as for outcome 23
Time Frame: as for outcome 23
Population: ITT/Evaluable population - Primary and expansion cohort combined
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Biliary Tract Cancer (BTC)
Number analyzed (Participants) | 43
Weeks | 58.9 [45.4 to 76.6]

25. Secondary Outcome: Overall Survival (OS) in the Adenocarcinoma of the Small Intestine (ASI) Cohort
Description: as for outcome 23
Time Frame: as for outcome 23
Population: ITT/Evaluable population - Primary analysis cohort
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Adenocarcinoma of the Small Intestine (ASI)
Number analyzed (Participants) | 3
Weeks | 94.6 [14.9 to NA] — Not estimable due to insufficient events observed

26. Secondary Outcome: Overall Survival (OS) in the Low Grade (WHO G1/G2) Glioma (LGG) Cohort
Description: as for outcome 23
Time Frame: as for outcome 23
Population: ITT/Evaluable population - Primary analysis cohort
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Low Grade (WHO G1/G2) Glioma (LGG)
Number analyzed (Participants) | 13
Weeks | NA [50.4 to NA] — Not estimable due to insufficient events observed

27. Secondary Outcome: Overall Survival (OS) in the High Grade (WHO G3/G4) Glioma (HGG) Cohort
Description: as for outcome 23
Time Frame: as for outcome 23
Population: ITT/Evaluable population - Primary and expansion cohort combined.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | High Grade (WHO G3/G4) Glioma (HGG)
Number analyzed (Participants) | 45
Weeks | 76.4 [41.1 to 139.9]

28. Secondary Outcome: Overall Survival (OS) in the Hairy Cell Leukemia (HCL) Cohort
Description: as for outcome 23
Time Frame: as for outcome 23
Population: ITT/Evaluable population - Primary and expansion cohort combined
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Hairy Cell Leukemia (HCL)
Number analyzed (Participants) | 55
Weeks | NA [NA to NA] — Not estimable due to insufficient events observed

29. Secondary Outcome: Overall Survival (OS) in the Multiple Myeloma (MM) Cohort
Description: as for outcome 23
Time Frame: as for outcome 23
Population: ITT/Evaluable population - Primary analysis cohort
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Multiple Myeloma (MM)
Number analyzed (Participants) | 10
Weeks | 147.3 [12.4 to 194.0]

30. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: The distribution of adverse events (AE) was done via the analysis of frequencies for treatment emergent Adverse Event (TEAEs) and Serious Adverse Event (TESAEs) through the monitoring of relevant clinical and laboratory safety parameters.
Time Frame: From study treatment start date till 30 days safety follow-up, assessed up to 92 months (cut-off date for end of study = 10-Dec-21)
Population: All-treated Subjects (ATS) population - Primary and expansion cohort combined
Measure: Count of Participants; unit: Participants
Arm/Group | Anaplastic Thyroid Cancer (ATC) | Biliary Tract Cancer (BTC) | Gastrointestinal Stromal Tumor (GIST) | Low Grade (WHO G1/G2) Glioma (LGG) | High Grade (WHO G3/G4) Glioma (HGG) | Adenocarcinoma of the Small Intestine (ASI) | Hairy Cell Leukemia (HCL) | Multiple Myeloma (MM)
Number analyzed (Participants) | 36 | 43 | 1 | 13 | 45 | 3 | 55 | 10
Participants
  Any AE | 36 | 43 | 1 | 12 | 42 | 3 | 55 | 9
  AEs related to study treatment | 27 | 42 | 1 | 12 | 37 | 3 | 52 | 7
  AEs leading to permanent discontinuation of any study treatment | 6 | 1 | 0 | 2 | 4 | 1 | 13 | 1
  AEs leading to dose reduction | 17 | 15 | 1 | 4 | 18 | 2 | 29 | 5
  AEs leading to dose interruption/delay | 19 | 24 | 1 | 6 | 18 | 2 | 40 | 6
  Any SAE | 20 | 17 | 1 | 3 | 16 | 0 | 32 | 4
  SAEs related to study treatment | 7 | 9 | 0 | 1 | 7 | 0 | 19 | 3
  Fatal SAEs | 3 | 2 | 0 | 0 | 1 | 0 | 3 | 0

31. Post Hoc Outcome: All Collected Deaths
Description: On-treatment deaths were collected from first dose of study medication to 30 days after study drug discontinuation, for a maximum duration of 85 months. Post-treatment survival follow-up deaths were collected from day 31 after last dose of first dose of study medication, up to 92 months. All deaths refer to the sum of on-treatment deaths and post-treatment survival follow-up deaths.
Time Frame: On-treatment deaths: Up to 85 months. Post-treatment survival follow-up deaths: Up to 92 months.
Population: All-treated Subjects (ATS) population - Primary and expansion cohort combined
Measure: Number; unit: Participants
Arm/Group | Anaplastic Thyroid Cancer (ATC) | Biliary Tract Cancer (BTC) | Gastrointestinal Stromal Tumor (GIST) | Low Grade (WHO G1/G2) Glioma (LGG) | High Grade (WHO G3/G4) Glioma (HGG) | Adenocarcinoma of the Small Intestine (ASI) | Hairy Cell Leukemia (HCL) | Multiple Myeloma (MM)
Number analyzed (Participants) | 36 | 43 | 1 | 13 | 45 | 3 | 55 | 10
Participants
  On-treatment deaths | 6 | 6 | 0 | 1 | 2 | 0 | 4 | 1
  Post-treatment survival follow-up deaths: number analyzed (Participants) | 30 | 37 | 1 | 12 | 43 | 3 | 51 | 9
  Post-treatment survival follow-up deaths | 18 | 28 | 1 | 3 | 26 | 3 | 4 | 8
  All deaths | 24 | 34 | 1 | 4 | 28 | 3 | 8 | 9

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 30 days, up to a maximum duration of approximately 85 months. Deaths were collected in the post treatment survival follow up period from 31 days after last dose of study medication until the end of the study, up to approximately 92 months. These are not considered Adverse Events.
Description: Any sign or symptom that occurred during the conduct of the trial and safety follow-up.
  Deaths in the post treatment survival follow-up period are not considered Adverse Events. The total number at risk in the post treatment survival follow-up period includes patients that entered the post treatment survival follow-up period.
Groups:
- Anaplastic Thyroid Cancer (ATC) (On-Treatment); Biliary Tract Cancer (BTC) (On-Treatment); Gastrointestinal Stromal Tumor (GIST) (On-Treatment); Low Grade (WHO G1/G2) Glioma (LGG) (On-Treatment); High Grade (WHO G3/G4) Glioma (HGG) (On-Treatment); Adenocarcinoma of the Small Intestine (ASI) (On-Treatment); Hairy Cell Leukemia (HCL) (On-Treatment); Multiple Myeloma (MM) (On-Treatment): All subjects enrolled received oral dabrafenib 150 mg bid in combination with oral trametinib 2 mg once daily. Subjects continued treatment until an unacceptable toxicity, disease progression, or death.
- Anaplastic Thyroid Cancer (ATC) (Post-treatment Survival Follow-up); Biliary Tract Cancer (BTC) (Post-treatment Survival Follow-up); Gastrointestinal Stromal Tumor (GIST) (Post-treatment Survival Follow-up); Low Grade (WHO G1/G2) Glioma (LGG) (Post-treatment Survival Follow-up); High Grade (WHO G3/G4) Glioma (HGG) (Post-treatment Survival Follow-up); Adenocarcinoma of the Small Intestine (ASI) (Post-treatment Survival Follow-up); Hairy Cell Leukemia (HCL) (Post-treatment Survival Follow-up); Multiple Myeloma (MM) (Post-treatment Survival Follow-up): Deaths collected in the post- treatment survival follow-up period (starting from day 31 post- treatment). No AEs were collected during this period.
Arm/Group | Anaplastic Thyroid Cancer (ATC) (On-Treatment) | Biliary Tract Cancer (BTC) (On-Treatment) | Gastrointestinal Stromal Tumor (GIST) (On-Treatment) | Low Grade (WHO G1/G2) Glioma (LGG) (On-Treatment) | High Grade (WHO G3/G4) Glioma (HGG) (On-Treatment) | Adenocarcinoma of the Small Intestine (ASI) (On-Treatment) | Hairy Cell Leukemia (HCL) (On-Treatment) | Multiple Myeloma (MM) (On-Treatment) | Anaplastic Thyroid Cancer (ATC) (Post-treatment Survival Follow-up) | Biliary Tract Cancer (BTC) (Post-treatment Survival Follow-up) | Gastrointestinal Stromal Tumor (GIST) (Post-treatment Survival Follow-up) | Low Grade (WHO G1/G2) Glioma (LGG) (Post-treatment Survival Follow-up) | High Grade (WHO G3/G4) Glioma (HGG) (Post-treatment Survival Follow-up) | Adenocarcinoma of the Small Intestine (ASI) (Post-treatment Survival Follow-up) | Hairy Cell Leukemia (HCL) (Post-treatment Survival Follow-up) | Multiple Myeloma (MM) (Post-treatment Survival Follow-up)
All-Cause Mortality (participants affected / at risk) | 6/36 | 6/43 | 0/1 | 1/13 | 2/45 | 0/3 | 4/55 | 1/10 | 18/30 | 28/37 | 1/1 | 3/12 | 26/43 | 3/3 | 4/51 | 8/9
Serious Adverse Events (participants affected / at risk) | 20/36 | 17/43 | 1/1 | 3/13 | 16/45 | 0/3 | 32/55 | 4/10 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 36/36 | 43/43 | 1/1 | 12/13 | 42/45 | 3/3 | 55/55 | 9/10 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anaplastic Thyroid Cancer (ATC) (On-Treatment) (N=36) | Biliary Tract Cancer (BTC) (On-Treatment) (N=43) | Gastrointestinal Stromal Tumor (GIST) (On-Treatment) (N=1) | Low Grade (WHO G1/G2) Glioma (LGG) (On-Treatment) (N=13) | High Grade (WHO G3/G4) Glioma (HGG) (On-Treatment) (N=45) | Adenocarcinoma of the Small Intestine (ASI) (On-Treatment) (N=3) | Hairy Cell Leukemia (HCL) (On-Treatment) (N=55) | Multiple Myeloma (MM) (On-Treatment) (N=10) | Anaplastic Thyroid Cancer (ATC) (Post-treatment Survival Follow-up) (N=0) | Biliary Tract Cancer (BTC) (Post-treatment Survival Follow-up) (N=0) | Gastrointestinal Stromal Tumor (GIST) (Post-treatment Survival Follow-up) (N=0) | Low Grade (WHO G1/G2) Glioma (LGG) (Post-treatment Survival Follow-up) (N=0) | High Grade (WHO G3/G4) Glioma (HGG) (Post-treatment Survival Follow-up) (N=0) | Adenocarcinoma of the Small Intestine (ASI) (Post-treatment Survival Follow-up) (N=0) | Hairy Cell Leukemia (HCL) (Post-treatment Survival Follow-up) (N=0) | Multiple Myeloma (MM) (Post-treatment Survival Follow-up) (N=0)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Leukopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Atrioventricular block (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Cardiac ventricular thrombosis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Conduction disorder (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Myocarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Stress cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Adrenocortical insufficiency acute (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Amaurosis fugax (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Haematochezia (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 3 | 0 | 2 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Fat necrosis (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Pyrexia (General disorders) | 1 | 9 | 0 | 1 | 1 | 0 | 10 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Cholangitis (Hepatobiliary disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Hepatic cytolysis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Bacterial diarrhoea (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Cervicitis human papilloma virus (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Enterobacter infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Gastroenteritis pseudomonas (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Lymph node tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Otitis media acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Parotitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Pelvic infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Pneumonia (Infections and infestations) | 8 | 1 | 0 | 0 | 0 | 0 | 4 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Pneumonia aspiration (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Pneumonia necrotising (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Sepsis (Infections and infestations) | 1 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Urinary tract infection (Infections and infestations) | 2 | 1 | 0 | 1 | 1 | 0 | 2 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Wound infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Ejection fraction decreased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Neutrophil count decreased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Transaminases increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Adenocarcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Aphasia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Central nervous system lesion (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Cerebral cyst (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Cerebral thrombosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Facial nerve disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Guillain-Barre syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Paralysis recurrent laryngeal nerve (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Device failure (Product Issues) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Hallucination (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Acute kidney injury (Renal and urinary disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Pulmonary haematoma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Aortic thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Thrombophlebitis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Anaplastic Thyroid Cancer (ATC) (On-Treatment) (N=36) | Biliary Tract Cancer (BTC) (On-Treatment) (N=43) | Gastrointestinal Stromal Tumor (GIST) (On-Treatment) (N=1) | Low Grade (WHO G1/G2) Glioma (LGG) (On-Treatment) (N=13) | High Grade (WHO G3/G4) Glioma (HGG) (On-Treatment) (N=45) | Adenocarcinoma of the Small Intestine (ASI) (On-Treatment) (N=3) | Hairy Cell Leukemia (HCL) (On-Treatment) (N=55) | Multiple Myeloma (MM) (On-Treatment) (N=10) | Anaplastic Thyroid Cancer (ATC) (Post-treatment Survival Follow-up) (N=0) | Biliary Tract Cancer (BTC) (Post-treatment Survival Follow-up) (N=0) | Gastrointestinal Stromal Tumor (GIST) (Post-treatment Survival Follow-up) (N=0) | Low Grade (WHO G1/G2) Glioma (LGG) (Post-treatment Survival Follow-up) (N=0) | High Grade (WHO G3/G4) Glioma (HGG) (Post-treatment Survival Follow-up) (N=0) | Adenocarcinoma of the Small Intestine (ASI) (Post-treatment Survival Follow-up) (N=0) | Hairy Cell Leukemia (HCL) (Post-treatment Survival Follow-up) (N=0) | Multiple Myeloma (MM) (Post-treatment Survival Follow-up) (N=0)
Anaemia (Blood and lymphatic system disorders) | 12 | 10 | 0 | 4 | 9 | 0 | 10 | 3 | NA | NA | NA | NA | NA | NA | NA | NA
Leukopenia (Blood and lymphatic system disorders) | 2 | 2 | 0 | 1 | 4 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 2 | 3 | 0 | 1 | 7 | 1 | 6 | 4 | NA | NA | NA | NA | NA | NA | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 7 | 0 | 1 | 4 | 0 | 3 | 3 | NA | NA | NA | NA | NA | NA | NA | NA
Atrial fibrillation (Cardiac disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 7 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Atrioventricular block first degree (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 13 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Tachycardia (Cardiac disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Ear pain (Ear and labyrinth disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 7 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 3 | 2 | 0 | 6 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Hypothyroidism (Endocrine disorders) | 4 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Cataract (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 4 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Diplopia (Eye disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Dry eye (Eye disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 5 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Eye pain (Eye disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Iritis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Macular oedema (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Papilloedema (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Photophobia (Eye disorders) | 1 | 0 | 0 | 1 | 3 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Saccadic eye movement (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Uveitis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Vision blurred (Eye disorders) | 1 | 1 | 0 | 2 | 5 | 0 | 14 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Visual impairment (Eye disorders) | 4 | 1 | 0 | 1 | 1 | 0 | 3 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 2 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 2 | 5 | 0 | 2 | 2 | 2 | 12 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 2 | 7 | 0 | 2 | 1 | 0 | 3 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Constipation (Gastrointestinal disorders) | 8 | 9 | 1 | 4 | 8 | 1 | 22 | 3 | NA | NA | NA | NA | NA | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | 7 | 14 | 0 | 4 | 5 | 1 | 19 | 3 | NA | NA | NA | NA | NA | NA | NA | NA
Dry mouth (Gastrointestinal disorders) | 5 | 8 | 0 | 2 | 3 | 0 | 8 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Dyspepsia (Gastrointestinal disorders) | 1 | 3 | 1 | 3 | 1 | 0 | 5 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Dysphagia (Gastrointestinal disorders) | 6 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 2 | 0 | 1 | 2 | 1 | 6 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Hyperaesthesia teeth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Nausea (Gastrointestinal disorders) | 12 | 18 | 1 | 7 | 14 | 0 | 27 | 5 | NA | NA | NA | NA | NA | NA | NA | NA
Noninfective gingivitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Oral pain (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Salivary gland mass (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Stomatitis (Gastrointestinal disorders) | 2 | 3 | 1 | 2 | 1 | 0 | 3 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Toothache (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 7 | 15 | 1 | 4 | 11 | 1 | 13 | 3 | NA | NA | NA | NA | NA | NA | NA | NA
Asthenia (General disorders) | 3 | 7 | 1 | 0 | 4 | 0 | 3 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Chills (General disorders) | 8 | 12 | 0 | 3 | 5 | 1 | 30 | 2 | NA | NA | NA | NA | NA | NA | NA | NA
Fatigue (General disorders) | 13 | 14 | 0 | 8 | 19 | 0 | 29 | 3 | NA | NA | NA | NA | NA | NA | NA | NA
Feeling cold (General disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Gait disturbance (General disorders) | 1 | 1 | 0 | 0 | 2 | 0 | 2 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Influenza like illness (General disorders) | 0 | 3 | 0 | 2 | 1 | 0 | 7 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Malaise (General disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 6 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Mucosal inflammation (General disorders) | 3 | 3 | 0 | 1 | 2 | 0 | 1 | 2 | NA | NA | NA | NA | NA | NA | NA | NA
Nodule (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Non-cardiac chest pain (General disorders) | 2 | 1 | 0 | 3 | 1 | 1 | 3 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Oedema (General disorders) | 1 | 3 | 0 | 0 | 2 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Oedema peripheral (General disorders) | 5 | 4 | 0 | 2 | 3 | 1 | 27 | 2 | NA | NA | NA | NA | NA | NA | NA | NA
Pain (General disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Peripheral swelling (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Pyrexia (General disorders) | 17 | 25 | 1 | 8 | 11 | 2 | 41 | 3 | NA | NA | NA | NA | NA | NA | NA | NA
Thirst (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Xerosis (General disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Sarcoidosis (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 5 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Conjunctivitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 8 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Folliculitis (Infections and infestations) | 1 | 2 | 0 | 1 | 3 | 0 | 2 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Fungal infection (Infections and infestations) | 2 | 0 | 0 | 0 | 1 | 0 | 4 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Herpes zoster (Infections and infestations) | 0 | 3 | 0 | 0 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | NA | NA | NA | NA | NA | NA | NA | NA
Nasopharyngitis (Infections and infestations) | 2 | 1 | 0 | 5 | 7 | 0 | 4 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Onychomycosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Oropharyngeal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Paronychia (Infections and infestations) | 0 | 1 | 0 | 1 | 3 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 0 | 6 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Rash pustular (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 5 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Sinusitis (Infections and infestations) | 2 | 1 | 0 | 1 | 1 | 0 | 4 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Skin candida (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Streptococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Tooth abscess (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Tooth infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 8 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Upper respiratory tract infection (Infections and infestations) | 3 | 1 | 0 | 0 | 2 | 0 | 15 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Urinary tract infection (Infections and infestations) | 2 | 2 | 0 | 1 | 6 | 1 | 8 | 2 | NA | NA | NA | NA | NA | NA | NA | NA
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 1 | 1 | 0 | 9 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Radiation associated pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Alanine aminotransferase increased (Investigations) | 4 | 7 | 0 | 3 | 9 | 0 | 18 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Aspartate aminotransferase increased (Investigations) | 5 | 11 | 0 | 4 | 9 | 0 | 21 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Blood alkaline phosphatase increased (Investigations) | 6 | 9 | 0 | 3 | 0 | 0 | 16 | 2 | NA | NA | NA | NA | NA | NA | NA | NA
Blood bilirubin increased (Investigations) | 0 | 3 | 0 | 0 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Blood creatine phosphokinase increased (Investigations) | 1 | 2 | 0 | 2 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Blood creatinine increased (Investigations) | 2 | 5 | 0 | 0 | 1 | 0 | 13 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Blood glucose increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0 | 1 | 2 | 0 | 4 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Blood oestrogen decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Blood testosterone decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Blood urea increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Blood uric acid increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
C-reactive protein increased (Investigations) | 0 | 1 | 0 | 0 | 2 | 0 | 2 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Ejection fraction decreased (Investigations) | 3 | 0 | 0 | 1 | 5 | 0 | 7 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Electrocardiogram QT prolonged (Investigations) | 3 | 0 | 0 | 1 | 1 | 0 | 5 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Gamma-glutamyltransferase increased (Investigations) | 3 | 12 | 0 | 1 | 2 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Glycosylated haemoglobin increased (Investigations) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Lipase increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Lymphocyte count decreased (Investigations) | 0 | 2 | 0 | 1 | 2 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Neutrophil count decreased (Investigations) | 3 | 4 | 0 | 3 | 8 | 0 | 2 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Neutrophil count increased (Investigations) | 2 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Platelet count decreased (Investigations) | 1 | 5 | 0 | 1 | 1 | 0 | 3 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Urine output decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Weight decreased (Investigations) | 4 | 3 | 0 | 1 | 0 | 1 | 3 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Weight increased (Investigations) | 1 | 4 | 0 | 3 | 1 | 1 | 2 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
White blood cell count decreased (Investigations) | 5 | 10 | 0 | 3 | 6 | 0 | 3 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 12 | 10 | 0 | 2 | 6 | 0 | 7 | 3 | NA | NA | NA | NA | NA | NA | NA | NA
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 8 | 0 | 2 | 4 | 0 | 25 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 4 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 1 | 0 | 0 | 3 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Hypoalbuminaemia (Metabolism and nutrition disorders) | 7 | 3 | 0 | 0 | 4 | 0 | 6 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Hypocalcaemia (Metabolism and nutrition disorders) | 5 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 3 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 4 | 0 | 0 | 2 | 0 | 3 | 2 | NA | NA | NA | NA | NA | NA | NA | NA
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 5 | 0 | 2 | 4 | 0 | 2 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 7 | 5 | 0 | 0 | 1 | 0 | 2 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 2 | 4 | 0 | 11 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 6 | 0 | 7 | 7 | 0 | 21 | 2 | NA | NA | NA | NA | NA | NA | NA | NA
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 4 | 0 | 3 | 3 | 0 | 13 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2 | 5 | 0 | 6 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 4 | 0 | 2 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 8 | 0 | 2 | 7 | 0 | 25 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 2 | 4 | 0 | 19 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | NA | NA | NA | NA | NA | NA | NA | NA
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1 | 0 | 13 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 0 | 2 | 0 | 2 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Dizziness (Nervous system disorders) | 7 | 1 | 0 | 2 | 5 | 0 | 20 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 5 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Epilepsy (Nervous system disorders) | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Facial paresis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Head discomfort (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Headache (Nervous system disorders) | 8 | 10 | 0 | 8 | 18 | 0 | 21 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 3 | 0 | 1 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
IIIrd nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Intercostal neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 3 | 1 | 0 | 2 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Neuropathy peripheral (Nervous system disorders) | 2 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Nystagmus (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Palatal palsy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Paraesthesia (Nervous system disorders) | 1 | 1 | 0 | 1 | 4 | 0 | 9 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Polyneuropathy (Nervous system disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Pyramidal tract syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
VIth nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Anxiety (Psychiatric disorders) | 1 | 3 | 0 | 1 | 0 | 0 | 4 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 3 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Depression (Psychiatric disorders) | 1 | 1 | 0 | 2 | 1 | 0 | 5 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Emotional disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Insomnia (Psychiatric disorders) | 5 | 6 | 0 | 2 | 2 | 1 | 9 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Libido decreased (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Mood swings (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Acute kidney injury (Renal and urinary disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Haematuria (Renal and urinary disorders) | 2 | 0 | 0 | 1 | 2 | 0 | 10 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 9 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Proteinuria (Renal and urinary disorders) | 2 | 1 | 0 | 3 | 1 | 0 | 2 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 10 | 0 | 3 | 8 | 0 | 30 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 7 | 0 | 0 | 2 | 0 | 13 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1 | 2 | 0 | 7 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 20 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2 | 1 | 0 | 11 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 0 | 0 | 0 | 9 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Acne (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 4 | 0 | 2 | 2 | NA | NA | NA | NA | NA | NA | NA | NA
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 4 | 0 | 2 | 5 | 0 | 22 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 4 | 0 | 5 | 2 | 1 | 17 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Eczema (Skin and subcutaneous tissue disorders) | 0 | 5 | 0 | 0 | 2 | 0 | 3 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Erythema (Skin and subcutaneous tissue disorders) | 1 | 5 | 0 | 3 | 1 | 0 | 5 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 8 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 4 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Night sweats (Skin and subcutaneous tissue disorders) | 3 | 3 | 0 | 3 | 1 | 2 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 4 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Piloerection (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 5 | 0 | 6 | 0 | 0 | 10 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 10 | 12 | 0 | 4 | 12 | 0 | 11 | 3 | NA | NA | NA | NA | NA | NA | NA | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 4 | 0 | 1 | 0 | 1 | 19 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Skin lesion (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Skin plaque (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Skin striae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Flushing (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 3 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Hypertension (Vascular disorders) | 1 | 6 | 0 | 2 | 2 | 1 | 8 | 1 | NA | NA | NA | NA | NA | NA | NA | NA
Hypotension (Vascular disorders) | 5 | 0 | 0 | 2 | 0 | 0 | 8 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA
Varicose vein (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/10/NCT02034110/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-10): https://cdn.clinicaltrials.gov/large-docs/10/NCT02034110/SAP_001.pdf